CLINICAL TRIAL: NCT03029663
Title: Complications of Transurethral Resection of the Bladder Tumour: A Prospective Analysis of Incidence and Predictive Factors
Brief Title: Complications of Transurethral Resection of the Bladder Tumour
Acronym: ComTUR
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: 12/2016
Record Dates: First submitted 2016-12-27; First posted 2017-01-24 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2017-01

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; postoperative complications
MeSH Terms: conditions — Urinary Bladder Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Transurethral resection of the bladder tumour

SUMMARY:
This is a prospective study enrolling consecutive patients who undergo transurethral resection of the bladder tumour (TURBT) aimed at determination of a safety of the procedure. Study end-points are incidence, severity and predictive factors of surgical complications. The study secondary aim is a validation of Clavien Dindo scoring system for reporting complication of TURBT.

ELIGIBILITY:
Inclusion Criteria:

* primary or recurrent bladder tumour
* informed consent to undergo the surgery

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing TURBT
Sampling Method: Non-Probability Sample
Enrollment: 983 (Actual)
Dates: Start 2016-12; Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Complications rate | 30 days postop

SECONDARY OUTCOMES:
Complications severity | 30 days postop
  Severity of surgical complications according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Dept. of Urology, Warsaw, Poland

REFERENCES:
- [Derived] Poletajew S, Krajewski W, Gajewska D, Sondka-Migdalska J, Borowik M, Buraczynski P, Dziegala M, Lykowski M, Przudzik M, Tukiendorf A, Wozniak R, Bar K, Jablonowski Z, Roslan M, Slojewski M, Zdrojowy R, Radziszewski P, Dziobek K. Prediction of the risk of surgical complications in patients undergoing monopolar transurethral resection of bladder tumour - a prospective multicentre observational study. Arch Med Sci. 2019 Oct 7;16(4):863-870. doi: 10.5114/aoms.2019.88430. eCollection 2020. PMID 32542089